CLINICAL TRIAL: NCT04405440
Title: Excessive Avoidance Behaviors in Anorexia Nervosa: the Role of Reward
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bram Vervliet (Other)
Responsible Party: Sponsor-Investigator, Bram Vervliet, Principal Investigator Prof. Dr. Bram Vervliet, KU Leuven
Organization: KU Leuven (Other)
Other Study IDs: S62060
Record Dates: First submitted 2019-11-28; First posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Eating Disorders; Anxiety; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anxiety Disorders; Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: The healthy control group will perform a well-validated avoidance (behavioral) task and will fill in some questionnaires about eating behaviors, emotions, and feelings.
  Interventions: Behavioral: Behavioral avoidance task
- Anorexia Nervosa patients: As the healthy controls, the participants of the anorexia nervosa group will perform the same behavioral task and will fill in the same questionnaires
  Interventions: Behavioral: Behavioral avoidance task

INTERVENTIONS:
Behavioral: Behavioral avoidance task — Behavioral task able to measure avoidance actions, US-expectancy, and reward-related indexes in different learning times

SUMMARY:
This study investigates excessive avoidance behaviors in patients with a diagnosis of Anorexia Nervosa (AN) compared to a healthy control group. The study further examines the role of reward (relief) as a putative factor in maintaining excessive avoidance behaviors in AN.

DETAILED DESCRIPTION:
Anorexia Nervosa (AN) is a life-threatening mental disease with a disappointing treatment outcome. Fear of weight gain and diet restrictions are considered the core symptoms of AN. Although from a diagnostic perspective AN is conceptualized as an eating-related disorder connected to an extremely low Body Mass Index (BMI) and body image distortion, AN might represent a specific phenotype of anxiety disorders characterized by tenacious avoidance behaviors, especially the restrictive subtype. To date, avoidance in AN is often investigated as a general personality trait (e.g. harm avoidance) but poorly examined in its behavioral form (which is life-threatening, such as food-avoidance). Hence, the investigators will perform a systematic investigation of excessive avoidance behaviors within a laboratory setting. Within a learning perspective, the investigators will investigate excessive avoidance in a group of 30 AN patients and 30 healthy volunteers. To achieve this, a well-validated avoidance paradigm will be used. Most critically, the investigators will examine whether patients with a diagnosis of anorexia nervosa show persistent avoidance behaviors compared to a control group. Additionally, the investigators will examine if, in the anorexia group, higher subjective relief to successful omissions of negative events during avoidance learning predicts persistent (excessive) avoidance behaviors after fear extinction.

ELIGIBILITY:
Inclusion Criteria:

* For the AN group, patients need to be physically strong and sufficiently emotionally stable
* For the healthy group, the investigators will recruit participants without a previous or current history of psychiatric, cardiovascular, neurological or other relevant disorder

Exclusion Criteria:

* For the AN group, the investigators will exclude patients who are insufficiently emotionally stable and/or physically weak to participate in the study as estimated by the treating physicians of the units on which the patients are admitted
* Insufficient verbal skills to understand the questionnaires and the computer task
* Participants who are pregnant or breastfeeding

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The anorexia patients are recruited from a primary care clinic. Healthy controls are recruited from the general population
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Button clicks during a red cue will be recorded as a measure of avoidance (binary response) | through study completion, an average of 1 year
  To investigate whether, compared to healthy controls, individuals with a diagnosis of anorexia nervosa show excessive avoidance behaviors (frequent clicking to prevent the aversive stimulus). Repeated measure ANOVA (analysis of variance) will be employed to evaluate differences between groups. If data will violate the assumption of normality, mixed or generalize methods will be used.
Relief pleasantness ratings (Visual Analog Scale, from neutral [0] to very pleasant [100]) | through study completion, an average of 1 year
  To investigate whether, compared to healthy controls, individuals with a diagnosis of anorexia nervosa show higher relief pleasantness during the omission of the aversive stimuli. The investigators will also test if such responses predict a return in avoidance behaviors (button click) after fear has been extinguished. Repeated measure ANOVA (analysis of variance) and multiple linear regressions will be employed to evaluate differences between groups. If data will violate the assumption of normality mixed or generalize methods will be used.

SECONDARY OUTCOMES:
US-Expectancy ratings (Likert scale from 0:no picture to 10:certainly a picture) | through study completion, an average of 1 year
  To investigate whether, compared to healthy controls, individuals with a diagnosis of anorexia nervosa show higher US-expectancies during both avoidance learning and fear extinction learning. Repeated measure ANOVA (analysis of variance) will be employed to evaluate differences between groups. If data will violate the assumption of normality mixed or generalize methods will be used.
Eating Disorders Inventory [EDI] | through study completion, an average of 1 year
  Higher scores at the EDI, and especially to the drive for thinness subscale, correlate with higher avoidance actions.
Distress Tolerance Scale [DTS] | through study completion, an average of 1 year
  Lower scores at the DTS correlate with higher relief and higher avoidance actions

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Claes, Prof. Dr., Principal Investigator — KU Leuven
Locations (2):
- Belgium (2):
  - Psychiatry | UZ Leuven campus Gasthuisberg, Leuven
  - University of KU Leuven, Faculteit Psychologie en Pedagogische Wetenschappen, Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaye WH, Bulik CM, Thornton L, Barbarich N, Masters K. Comorbidity of anxiety disorders with anorexia and bulimia nervosa. Am J Psychiatry. 2004 Dec;161(12):2215-21. doi: 10.1176/appi.ajp.161.12.2215. PMID 15569892
- [Background] Godart NT, Flament MF, Lecrubier Y, Jeammet P. Anxiety disorders in anorexia nervosa and bulimia nervosa: co-morbidity and chronology of appearance. Eur Psychiatry. 2000 Feb;15(1):38-45. doi: 10.1016/s0924-9338(00)00212-1. PMID 10713801
- [Background] Koskina A, Campbell IC, Schmidt U. Exposure therapy in eating disorders revisited. Neurosci Biobehav Rev. 2013 Feb;37(2):193-208. doi: 10.1016/j.neubiorev.2012.11.010. Epub 2012 Nov 29. PMID 23201859
- [Background] Murray SB, Loeb KL, Le Grange D. Dissecting the Core Fear in Anorexia Nervosa: Can We Optimize Treatment Mechanisms? JAMA Psychiatry. 2016 Sep 1;73(9):891-2. doi: 10.1001/jamapsychiatry.2016.1623. No abstract available. PMID 27463780
- [Background] Murray SB, Strober M, Craske MG, Griffiths S, Levinson CA, Strigo IA. Fear as a translational mechanism in the psychopathology of anorexia nervosa. Neurosci Biobehav Rev. 2018 Dec;95:383-395. doi: 10.1016/j.neubiorev.2018.10.013. Epub 2018 Oct 28. PMID 30392878
- [Background] Wierenga CE, Bischoff-Grethe A, Melrose AJ, Irvine Z, Torres L, Bailer UF, Simmons A, Fudge JL, McClure SM, Ely A, Kaye WH. Hunger does not motivate reward in women remitted from anorexia nervosa. Biol Psychiatry. 2015 Apr 1;77(7):642-52. doi: 10.1016/j.biopsych.2014.09.024. Epub 2014 Oct 22. PMID 25481622
- [Background] Park RJ, Godier LR, Cowdrey FA. Hungry for reward: How can neuroscience inform the development of treatment for Anorexia Nervosa? Behav Res Ther. 2014 Nov;62:47-59. doi: 10.1016/j.brat.2014.07.007. Epub 2014 Jul 26. PMID 25151600